CLINICAL TRIAL: NCT04765514
Title: A Randomized Controlled Trial of Chemo-Radiotherapy Versus Biomarker-Guided Therapy for Elderly and Frail Patients With Newly Diagnosed Glioblastoma
Brief Title: Chemoradiotherapy Versus Biomarker-Guided Therapy for Elderly and Frail GBM Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0012
Record Dates: First submitted 2021-01-12; First posted 2021-02-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Arm: TMZ with concurrent RT (combined modality arm) (Active Comparator): Patients will receive a total of 21 days of Temozolomide (TMZ), with 15 days of TMZ administered daily with concurrent RT. TMZ will be delivered at a dose of 75 mg/m2, given daily with RT for 15 days, one hour before each session of RT.
  After a 4-week break, patients will receive six cycles of adjuvant TMZ according to the standard 5-day schedule (days 1-5) every 28 days, up to 6 cycles as tolerated by the patient. The dose will be 150 mg/m2 for the first cycle and increased to 200 mg/m2 beginning with the second cycle, so long as there are no hematologic adverse events, intractable nausea or fatigue.
  Interventions: Combination Product: Chemo-Radiotherapy consisting of 40 Gy in 15 daily fractions with concurrent temozolomide.
- Biomarker based treatment (Experimental): MGMT (+) Temozolomide monotherapy: Patients will receive Temozolomide (TMZ) at a dose of 75 mg/m2 daily for 21 consecutive days. This will be followed by six cycles of TMZ according to the standard 5-day schedule (days 1-5) every 28 days. The dose will be 150 mg/m2 for the first cycle and increased to 200 mg/m2 beginning with the second cycle, so long as there are no hematologic adverse events. Dose will be determined using body surface area (BSA) calculation.
  MGMT methylation (-) RT monotherapy: Participants will receive radiation treatment with 40Gy / 15 fractions over a period of 21 days (3 weeks).
  Interventions: Other: Biomarker based treatment (Temozolomide monotherapy or Radiotherapy monotherapy)

INTERVENTIONS:
Other: Biomarker based treatment (Temozolomide monotherapy or Radiotherapy monotherapy) — Temozolomide or Radiotherapy
  Arms: Biomarker based treatment
Combination Product: Chemo-Radiotherapy consisting of 40 Gy in 15 daily fractions with concurrent temozolomide. — Temozolomide will be administered at a dose of 75 mg/m2 daily for a total of 21 days. This will be followed by adjuvant temozolomide (150-200 mg/m2 daily for 5 day
  Arms: Standard Arm: TMZ with concurrent RT (combined modality arm)

SUMMARY:
Currently, the optimal treatment regimen for elderly Glioblastoma (GBM) patients with poor performance status (PS) is unknown. Based on data for elderly GBM patients and the limited data for patients with poor PS, hypofractionated RT or a short course of Temozolomide (TMZ) may provide survival benefit without the added toxicity and inconvenience of a more protracted treatment regimen.

In particular, treatment with RT or TMZ monotherapy on the basis of methylated O6 - methyl guanine - DNA methyltransferase (MGMT) promoter methylation status, followed by the alternative therapy at progression, may provide a safe and effective treatment regimen for patients with poor PS.

The hypothesis of this trial is that in elderly GBM patients with poor performance status (age ≥ 65 years and KPS 50-70), a biomarker-guided approach to therapy results in non-inferior overall survival compared to combined TMZ/RT.

Specifically, biomarker-guided therapy will consist of TMZ monotherapy for patients with a methylated MGMT promoter, and hypofractionated RT (40 Gy in 15 fractions) for patients with a non-methylated MGMT promoter.

It is hypothesized that biomarker-guided therapy will result in non-inferior progression-free survival, reduced toxicity and increased cost-effectiveness compared to combined chemoradiotherapy.

Primary objective:

• To compare overall survival of standard vs biomarker-guided therapy in elderly and frail patients with newly diagnosed GBM.

Secondary objective:

* To evaluate progression-free survival following treatment in both arms.
* To evaluate adverse events according to CTCAE criteria in both arms.
* To evaluate health-related quality-of-life as assessed by MoCA and EORTC QLQ-C30/QLQ-BN20 questionnaires in both arms.
* To evaluate cost-effectiveness of standard vs biomarker-guided therapy

Methods:

Patients will be randomized to two treatment groups in a 1:1 ratio. Standard Arm: TMZ with concurrent RT (combined modality arm) Patients will receive 15 days of TMZ daily with concurrent RT. TMZ will be delivered at a dose of 75 mg/m2, given daily with RT. TMZ will be administered 1 hour before each session of RT.

After a 4-week break, patients will receive six cycles of adjuvant TMZ according to the standard 5-day schedule (days 1-5) every 28 days, up to 6 cycles as tolerated by the patient. The dose will be 150 mg/m2 for the first cycle and increased to 200 mg/m2 beginning with the second cycle, so long as there are no hematologic adverse events, intractable nausea or fatigue.

Investigational Arm: Biomarker based treatment MGMT (+): TMZ monotherapy Patients will receive TMZ at a dose of 75 mg/m2 daily for 15 days on weekdays (Monday through Friday). This will be followed by six cycles of TMZ according to the standard 5-day schedule (days 1-5) every 28 days. The dose will be 150 mg/m2 for the first cycle and increased to 200 mg/m2 beginning with the second cycle, so long as there are no hematologic adverse events. Dose will be determined using the body surface area (BSA) calculation.

MGMT methylation (-): No TMZ will be given. Participants will receive radiation treatment with 40Gy / 15 fractions over a period of 21 days (3 weeks).

Upon treatment completion, participants will be followed by every 3 months for 2 years and every 6 months for years 3-5. Response and progression will be evaluated using the new international criteria proposed by the Response Assessment in Neuro-Oncology working group (RANO).

ELIGIBILITY:
Inclusion Criteria:

1. Newly-diagnosed, histologically proven, intracranial glioblastoma with maximal safe resection. Biopsy alone is expected if resection is not possible. MGMT promoter methylation status must be tested for all patients.
2. History and physical examination, including neurological examination, within 14 days prior to randomization.
3. Age ≥ 65 & KPS of 60 - 70
4. Stable or decreasing dose of corticosteroids for at least 14 days prior to randomization.
5. Laboratory evaluation within 7 days prior to randomization, with adequate function as defined below:

   1. ANC ≥ 1.5 x 109/L
   2. Platelets ≥ 100 x 109/L
   3. Estimated Glomerular Filtration Rate (eGFR) > 59
   4. Total serum bilirubin ≤ 30 umol/L (ie ≤ 1.5 times ULN)
   5. ALT < 150 U/L (ie < 3 times ULN)
   6. AST < 120 U/L (ie < 3 times ULN)
   7. Alkaline phosphatase < 390 U/L (ie < 3 times ULN)
6. Patients must sign a study-specific informed consent prior to study registration.
7. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 6 months after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

   Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
   1. This will apply for male patients only and their female partner if of child bearing potential.
   2. Effective contraception should also be used by male patients taking temozolomide. Men being treated with temozolomide are advised not to father a child during or up to 6 months after discontinuation of treatment (male patients).
8. Male patients should agree to not donate sperm during the study treatment and for six months post treatment completion.

Exclusion Criteria:

1. Recurrent malignant gliomas
2. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years.
3. Prior head or neck RT (except for T1 glottic cancer), or systemic therapy precluding delivery of concurrent and adjuvant temozolomide
4. Treatment with any other therapeutic clinical protocol within 30 days prior to study registration or during participation in the study.
5. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization
   2. Transmural myocardial infarction within the last 6 months
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study registration
   4. Any severe, active co-morbidity precluding delivery of temozolomide.
   5. History of hypersensitivity reaction to temozolomide components or to dacarbazine.
   6. Active HBV infection

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Through study completion, an average of 2 years.
  Time between randomization and death due to any cause. Patients without an event will be censored the last time they were known to be alive.

SECONDARY OUTCOMES:
Progression-free survival | Median, 6-month, 1-year, and 2-year rates will be measured.
  Time between randomization and radiographic progression based on RANO criteria or death due to any cause. Patients without an event will be censored at the date of last follow-up for progression.
Frequency of Adverse Events related to the treatment administered | From screening until one month post adjuvant treatment.
  Adverse events related to the treatment(s) administered will be recorded from screening until one month post adjuvant treatment. Adverse events will be assessed according to NCI CTCAE version 4.0 criteria.
Health Related Quality of Life (EORTC QLQ-C30) | Throughout study completion, up to 5 years.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Health Related Quality of Life (EORTC QLQ-BN20) | Throughout study completion, up to 5 years.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Cost effectiveness | Upon study completion, an average of 5 years
  Assessed by the incremental cost-effectiveness ratio (ICER), calculated as: Cost per life-year gained = (Difference in direct costs between biomarker-guided therapy and chemoradiotherapy) ÷ (Difference in life-years gained between biomarker-guided therapy and chemoradiotherapy). The direct unit costs of TMZ and associated laboratory testing, RT, and costs associated with any grade 3-4 adverse events (eg hospitalization) will be included.
Cognitive and mental function | Throughout study completion, up to 5 years.
  Assessed by Montreal Cognitive Assessment (MoCA). This assessment was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No